CLINICAL TRIAL: NCT01745393
Title: Pediatrician Advice, Family Counseling & SHS Reduction for Underserved Children
Brief Title: Kids Safe and Smokefree (KiSS)
Acronym: KiSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Children's Hospital of Philadelphia (Other); St. Christopher's Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01CA158361 (NIH)
Record Dates: First submitted 2012-11-12; First posted 2012-12-10 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Second Hand Tobacco Smoke; Nicotine Dependence
Keywords: Smoking Cessation; Secondhand Smoke; Passive Smoking; Cotinine; Nicotine Replacement Products
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinic Quality Improvement + Behavioral Counseling (Experimental): This multilevel intervention includes advice and a referral from a pediatrician, behavioral counseling by study staff, and community systems navigation, all designed to reduce pediatric secondhand smoke exposure. Over the course of 12 weeks participants receive a home visit designed to orient them to the program and trained health counselors provide multiple individualized phone counseling sessions designed to build coping skills, urge management skills, and self-efficacy. Counseling also includes assistance with goal setting and navigation of local resources.
  Interventions: Behavioral: Clinic Quality Improvement + Behavioral Counseling
- Clinic Quality Improvement + Attention Control (Active Comparator): The attention control intervention parallels the format of the experimental group but focuses on family nutrition information. The intervention includes a home visit to orient the participant to the program and multiple phone counseling sessions conducted by a trained health counselor.
  Interventions: Behavioral: Clinic Quality Improvement + Attention Control

INTERVENTIONS:
Behavioral: Clinic Quality Improvement + Behavioral Counseling
  Arms: Clinic Quality Improvement + Behavioral Counseling
Behavioral: Clinic Quality Improvement + Attention Control
  Arms: Clinic Quality Improvement + Attention Control

SUMMARY:
The study's primary aim is to test the hypothesis that an intervention integrating pediatric clinic-level quality improvement with home-level behavioral counseling (CQI+BC) will result in greater reductions in child cotinine (a biomarker of secondhand smoke exposure) and reported cigarettes exposed/day than a clinic-level quality improvement plus attention control intervention (CQI+A). A secondary aim is to test the hypothesis that relative to CQI+A, CQI+BC will result in higher cotinine-verified, 7-day point prevalence quit rate among parents.

DETAILED DESCRIPTION:
Child secondhand smoke exposure (SHSe) is a significant public health problem that has been linked to asthma, acute respiratory illnesses, otitis, and SIDS, and is associated with increased risk of cancers, cardiovascular disease, and behavior problems. This project will test the effectiveness of a comprehensive multilevel intervention to reduce young children's SHSe in minority and medically underserved communities known to have the highest SHSe-related morbidity and mortality risk. First, we will provide a clinic-level quality improvement (CQI) intervention to improve the care of pediatric patients with SHSe in four pediatric clinics in North and West Philadelphia. We will then randomize eligible parents visiting the CQI clinics into either a home-level behavioral counseling intervention (CQI+BC) or a home-level attention control intervention (CQI+A). In addition to clinic-level intervention, CQI+BC provides personalized, behavioral counseling with intensive skills training and support where SHSe occurs (in the home), as well as systems navigation to facilitate access to and effective use of reimbursable nicotine replacement therapy and smoking cessation medication. Participants will complete assessments at pre-treatment, 3-month end of treatment, and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* English-speaking
* parent or legal guardian of child under 11 years old who lives with him/her
* daily smoker

Exclusion Criteria:

* non-nicotine drug dependence
* psychiatric disturbance (bipolar, schizophrenia, psychosis)
* pregnant
* inadequate health literacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2012-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Collins, PhD, Principal Investigator — Temple University; Stephen Lepore, PhD, Principal Investigator — Temple University
Locations (4):
- United States (4):
  - Children's Hospital of Philadephia, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Temple University Hospital System, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Lepore SJ, Winickoff JP, Moughan B, Bryant-Stephens TC, Taylor DR, Fleece D, Davey A, Nair US, Godfrey M, Collins BN. Kids Safe and Smokefree (KiSS): a randomized controlled trial of a multilevel intervention to reduce secondhand tobacco smoke exposure in children. BMC Public Health. 2013 Aug 30;13:792. doi: 10.1186/1471-2458-13-792. PMID 23987302
- [Result] Collins BN, Lepore SJ, Winickoff JP, Nair US, Moughan B, Bryant-Stephens T, Davey A, Taylor D, Fleece D, Godfrey M. An Office-Initiated Multilevel Intervention for Tobacco Smoke Exposure: A Randomized Trial. Pediatrics. 2018 Jan;141(Suppl 1):S75-S86. doi: 10.1542/peds.2017-1026K. PMID 29292308
- [Derived] Chin SM, Lepore SJ, Collins BN, Dumenci L, Rincon MA. Validation and Psychometric Properties of the Tobacco Urge Management Scale (TUMS). Int J Environ Res Public Health. 2023 Apr 10;20(8):5453. doi: 10.3390/ijerph20085453. PMID 37107735
- [Derived] Collins BN, Lepore SJ, Winickoff JP, Sosnowski DW. Parents' Self-efficacy for Tobacco Exposure Protection and Smoking Abstinence Mediate Treatment Effects on Child Cotinine at 12-Month Follow-up: Mediation Results from the Kids Safe and Smokefree Trial. Nicotine Tob Res. 2020 Oct 29;22(11):1981-1988. doi: 10.1093/ntr/ntz175. PMID 31536116
- [Derived] Lepore SJ, Collins BN, Sosnowski DW. Self-efficacy as a pathway to long-term smoking cessation among low-income parents in the multilevel Kids Safe and Smokefree intervention. Drug Alcohol Depend. 2019 Nov 1;204:107496. doi: 10.1016/j.drugalcdep.2019.05.027. Epub 2019 Aug 24. PMID 31499240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-assignment clinic-level intervention and referral (recruitment): Across five pediatric primary care clinics in Philadelphia's three largest pediatric health systems (Temple University, Drexel University, and Children's Hospital of Philadelphia), 334 providers conducted the Ask, Advise, Refer clinic-level treatment implemented for this study.
Pre-assignment Details: Providers referred 2949 parents to the trial: 1280 were not eligible, 598 declined participation, 702 could not be contacted. Of 369 at baseline, 369 completed self-report assessments; 42 did not complete the pre-randomization home-visit child urine (cotinine) pick-up. Thus, 327 participants were randomized between the two treatment conditions.
Groups:
- Clinic Quality Improvement + Behavioral Counseling: This multilevel intervention includes advice and a referral from a pediatrician, behavioral counseling by study staff, and community systems navigation, all designed to reduce pediatric secondhand smoke exposure. Over the course of 12 weeks participants receive a home visit designed to orient them to the program and trained health counselors provide multiple individualized phone counseling sessions designed to build coping skills, urge management skills, and self-efficacy. Counseling also includes assistance with goal setting and navigation of local resources.
  Clinic Quality Improvement + Behavioral Counseling
- Clinic Quality Improvement + Attention Control: The attention control intervention parallels the format of the experimental group but focuses on family nutrition information. The intervention includes a home visit to orient the participant to the program and multiple phone counseling sessions conducted by a trained health counselor.
  Clinic Quality Improvement + Attention Control
Period: Treatment to End-of-treatment Assessment
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control
Started | 163 | 164
Received Treatment | 147 (Behavioral counseling = TSE-reduction and cessation counseling via telephone) | 144 (Attention control = nutrition education via telephone)
Completed (completed end-of-treatment assessments) | 142 | 156
Not Completed | 21 | 8
Not completed — Lost to Follow-up | 20 | 8
Not completed — Withdrawal by Subject | 1 | 0
Period: 12-month Follow-up
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control
Started | 142 | 156
Completed | 136 | 151
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control | Total
Number analyzed (Participants) | 163 | 164 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.74 (7.94) | 33.88 (9.20) | 33.31 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 133 | 273
  Male | 23 | 31 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 134 | 138 | 272
  White | 9 | 9 | 18
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 163 | 164 | 327
married, living with partner [Count of Participants; unit: Participants] | 71 | 63 | 134
less than high school education [Count of Participants; unit: Participants] | 43 | 46 | 89
income below poverty level [Count of Participants; unit: Participants] | 128 | 129 | 257
child age [Mean (Standard Deviation); unit: months] — measured in months
  months | 64.53 (31.59) | 64.04 (33.87) | 64.29 (32.70)
parents' cigarettes per day smoked [Mean (Standard Deviation); unit: cigarettes smoked per day] | 12.18 (8.92) | 10.72 (5.84) | 11.45 (7.56)
child (log) cotinine [Mean (Standard Deviation); unit: log transformed ng/mL] | 1.17 (0.53) | 1.24 (0.50) | 1.21 (0.52)

OUTCOME MEASURES:

1. Primary Outcome: Child Urine Cotinine
Description: Child urine cotinine is a biomarker for assessing second-hand smoke exposure. We anticipate the CQI+BC treatment group will experience a greater reduction in child urine cotinine over time than the CQI+A control group.
Time Frame: up to 12 months
Population: The fewer number of units analyzed compared to participants analyzed relates to completion of telephone assessments for all participants, but inability to collect 5 urine samples in the Behavioral Counseling group and 2 urine samples in the Attention Control group at the post-phone assessment urine pickup at participants' homes.
Measure: Mean (Standard Deviation); unit: log transformed ng/mL
Units Other Than Participants: urine cotinine samples
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control
Number analyzed (Participants) | 136 | 151
Number analyzed (urine cotinine samples) | 131 | 149
log transformed ng/mL | 0.892 (0.65) | 0.891 (0.58)

2. Primary Outcome: Parent-reported Second-hand Smoke Exposure in Cigarettes Per Day From All Sources
Description: Parental report of cigarettes child is exposed to each day in the home and car by all sources during the 7 days prior to assessment. We anticipate the CQI+BC treatment group will report greater reductions in second-hand smoke exposure over time than the CQI+A control group.
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: cigarettes exposed per day
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control
Number analyzed (Participants) | 136 | 151
cigarettes exposed per day | 3.8 (5.52) | 3.04 (3.84)

3. Secondary Outcome: Parent-reported Cotinine-verified 7-day Point Prevalence Abstinence
Description: When a participant reports smoking abstinence, we will bioverify their smoking status.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control
Number analyzed (Participants) | 132 | 149
Participants | 20 | 10

ADVERSE EVENTS:
Time Frame: 1 year (from enrollment to 12-month follow-up assessment)
Description: There were no serious adverse events anticipated in this behavioral counseling trial designed to help parents reduce children's exposure to secondhand smoke and help parents quit smoking. However, we did track adverse events.
Arm/Group | Clinic Quality Improvement + Behavioral Counseling | Clinic Quality Improvement + Attention Control
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/164
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/164
Other Adverse Events (participants affected / at risk) | 0/163 | 0/164

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No